CLINICAL TRIAL: NCT01929213
Title: A Randomized, Open-label, Multiple Dose, Three-treatment, Three-period, Six-sequence Williams Design to Investigate the Pharmacokinetic Drug Interaction Between Udenafil and Bosentan After Oral Administration in Healthy Volunteers
Brief Title: Clinical Trial to Investigate the Pharmacokinetic Drug Interaction Between Udenafil and Bosentan After Oral Administration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA8159_PAH_DI
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — udenafil; Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Udenafil (Experimental)
  Interventions: Drug: Udenafil
- Bosentan (Experimental)
  Interventions: Drug: Bosentan
- Udenafil/Bosentan (Experimental)
  Interventions: Drug: Udenafil/Bosentan

INTERVENTIONS:
Drug: Udenafil — Udenafil is administered
  Arms: Udenafil
Drug: Bosentan — Bosentan is administered
  Arms: Bosentan
Drug: Udenafil/Bosentan — Udenafil and Bosentan are administered
  Arms: Udenafil/Bosentan

SUMMARY:
This study is designed to investigate the pharmacokinetic drug interaction and safety after oral administration of Udenafil(DA-8159) and Bosentan in healthy volunteers.

Design: Randomized, open-label, multiple-dose, three-treatment, three-period, six-sequence, Williams design

Investigational Product: Udenafil, Bosentan

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers between the ages of 20 to 45 years old within the range of BMI between 18.5 and 25(Body Mass Index)
* having neither congenital/chronic diseases nor pathological symptoms/findings as results of medical examination
* doctor determines to be suitable as subjects within 4 weeks ago before administration

Exclusion Criteria:

* Hypersensitivity(or history of hypersensitivity) to Udenafil, Bosentan and PDE5 inhibitors
* Active Liver Diseases or exceed 1.25 times the normal range of AST, ALT
* Gastrointestinal diseases or surgeries that affect absorption of drug
* Excessive drinking(exceed 210g/week) and excessive caffeine(exceed 5cups/day)
* Smoking over 10 cigarettes per day
* pregnant or nursing female volunteers

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Udenafil, Bosentan C max,ss | Blood gathering point: 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12h of D1, D15, D29(if Udenafil adminstrated alone), 0 h of D7, D21, D35, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 h of D8, D22, D36
Udenafil, Bosentan AUC tau,ss | Blood gathering point: 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12h of D1, D15, D29(if Udenafil adminstrated alone), 0 h of D7, D21, D35, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36 h of D8, D22, D36

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital Clinical Trial Center, Seoul, South Korea